CLINICAL TRIAL: NCT04426045
Title: Pericapsular Nerve Group (PENG) Block Versus Supra-inguinal Fascia Iliaca Compartment Block for Pain Management After Total Hip Arthroplasty: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4-2020-0417
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Total Hip Arthroplasty; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pericapsular nerve group block (Experimental): Participants receiving pericapsular nerve group block
  Interventions: Procedure: Pericapsular nerve group block
- Supra-inguinal fascia iliaca compartment block (Active Comparator): Participants receiving supra-inguinal fascia iliaca compartment block
  Interventions: Procedure: Supra-inguinal fascia iliaca compartment block

INTERVENTIONS:
Procedure: Pericapsular nerve group block — A curvilinear 2-5MHz ultrasound probe will be initially placed in a transverse plane over the anterior superior iliac spine and then aligned with the pubic ramus by rotating the probe counterclockwise approximately 45 degrees. In this view, the iliopubic eminence, the iliopsoas muscle and tendon, the femoral artery, and pectineus muscle will be observed. A 22-gauge, 80-mm needle will be inserted from lateral to medial in an in-plane approach to place the tip in the musculofascial plane between the psoas tendon anteriorly and the pubic ramus posteriorly. A total volume of 20 ml of ropivacaine 0.2% will be injected.
  Other Names: PENG block
  Arms: Pericapsular nerve group block
Procedure: Supra-inguinal fascia iliaca compartment block — A linear 6-13-MHz ultrasound probe will be placed in the sagittal plane to obtain an image of the anterior superior iliac spine. The fascia iliaca and sartorius, iliopsoas, and oblique internal muscles will be identified by sliding the probe medially. After identifying the "bow-tie sign" formed by the muscle fascias, a 22-gauge, 80-mm needle will be introduced 1 cm cephalad to the inguinal ligament. Using an in-plane approach, the fascia iliaca will be penetrated and hydrodissected, separating the fascia iliaca from the iliac muscle. A total volume of 30 ml of ropivacaine 0.2% will be injected.
  Other Names: Supra-inguinal FICB
  Arms: Supra-inguinal fascia iliaca compartment block

SUMMARY:
Adequate pain control after total hip arthroplasty is crucial for early ambulation and patient satisfaction. The supra-inguinal fascia iliaca compartment block has been described as a promising technique for primary total hip arthroplasty. However, one of the concerns with supra-inguinal fascia iliaca compartment block is still the potential for quadriceps weakness that might delay ambulation. The pericapsular nerve group (PENG) block has been recently introduced a new technique for blockade of the articular branches of the femoral, obturator and accessory obturator nerves. PENG block is possible to provide sufficient analgesia and preserve lower limb muscle strength. The investigators will compare ultrasound-guided supra-inguinal fascia iliaca compartment block with PENG block in patients undergoing total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19 years old or older, with American Society of Anesthesiologists Physical Status 1-3
* scheduled for elective unilateral total hip arthroplasty

Exclusion Criteria:

* Allergy or intolerance to any of the drugs used in the study
* Hepatic or renal insufficiency
* Opioid dependency
* Coagulopathy
* Pre-existing neurologic or anatomic deficits in the lower extremities
* Severe psychiatric illness

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2021-06-06 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale pain score | 1 hour after the surgery
  Pain intensity at rest and during 45-degree passive flexion of the hip with the ipsilateral knee flexed naturally will be evaluated by an 11-point numeric rating scale (NRS: 0 = no pain, 10 = worst imaginable pain)
Numeric rating scale pain score | 6 hours after the surgery
  Pain intensity at rest and during 45-degree passive flexion of the hip with the ipsilateral knee flexed naturally will be evaluated by an 11-point numeric rating scale (NRS: 0 = no pain, 10 = worst imaginable pain)
Numeric rating scale pain score | 24 hours after the surgery
  Pain intensity at rest and during 45-degree passive flexion of the hip with the ipsilateral knee flexed naturally will be evaluated by an 11-point numeric rating scale (NRS: 0 = no pain, 10 = worst imaginable pain)
Numeric rating scale pain score | 36 hours after the surgery
  Pain intensity at rest and during 45-degree passive flexion of the hip with the ipsilateral knee flexed naturally will be evaluated by an 11-point numeric rating scale (NRS: 0 = no pain, 10 = worst imaginable pain)
Numeric rating scale pain score | 48 hours after the surgery
  Pain intensity at rest and during 45-degree passive flexion of the hip with the ipsilateral knee flexed naturally will be evaluated by an 11-point numeric rating scale (NRS: 0 = no pain, 10 = worst imaginable pain)

SECONDARY OUTCOMES:
Quadriceps muscle strength | baseline
  Quadriceps muscle strength will be measured by the dynamometer
Quadriceps muscle strength | at 6 hours postoperatively
  Quadriceps muscle strength will be measured by the dynamometer
Quadriceps muscle strength | at 24 hours postoperatively
  Quadriceps muscle strength will be measured by the dynamometer
Quadriceps muscle strength | at 36 hours postoperatively
  Quadriceps muscle strength will be measured by the dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No